CLINICAL TRIAL: NCT06509516
Title: Quasi-experimental Study Protocol to Measure the Effect of Modified Sleeper-Stretch on the Elasticity of the Posterior and Posteroinferior Glenohumeral Capsule by Means of Shear Wave Elastography in Adult Population
Brief Title: Effect of the Modified Sleeper-Stretch on the Elasticity of the Posterior and Posteroinferior Glenohumeral Capsule
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Esteban Ramírez Llano, Physical Therapist, University of Alcala
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/3/066
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Pain; Shoulder Pain Chronic
Keywords: Modified Sleeper-Stretch; Shear Wave Elastography; Posterior Capsule; GIRD
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The same intervention, a programme of the Modified Sleeper-Stretch, will be applied on two different groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder pain history (Experimental): Execution of the Modified Sleeper-Stretch three times, for thirty seconds each time, with thirty seconds between stretches, daily, for twenty-eight days. The stretch will be applied on the shoulder with history of shoulder pain.
  Interventions: Other: Modified Sleeper-Stretch
- No history of shoulder pain (Experimental): Execution of the Modified Sleeper-Stretch three times, for thirty seconds each time, with thirty seconds between stretches, daily, for twenty-eight days. The stretch will be applied on a shoulder randomly assigned.
  Interventions: Other: Modified Sleeper-Stretch

INTERVENTIONS:
Other: Modified Sleeper-Stretch — Self-administered stretch in which the individual remains side-lying on the upper limb to be stretched, keeping the scapula stabilized by his/her own weight, and rolls the trunk 20-30º posteriorly, maintaining a 90º flexion in the shoulder and elbow. Using the opposite hand over the forearm of the limb to be stretched, the individual passively brings the shoulder to maximum internal rotation.

SUMMARY:
The goal of this quasi-experimental study is to determine the effect of the self-administered Modified Sleeper-Stretch on the elasticity of the posterior and posteroinferior glenohumeral capsule in adult individuals of both genders who either have clinical history of non-specific shoulder pain in a single shoulder or have no history of shoulder pain at all, being the assessment made by means of shear wave elastography. The main hypothesis it aims to confirm is:

• A soft tissue stretching program, using the Modified Sleeper-Stretch, aimed at general adult population with history of nonspecific shoulder pain that has occurred with glenohumeral internal rotation deficit improves the elasticity of the posterior and posteroinferior glenohumeral capsules, showing no significant effect on general adult population without history of shoulder pain.

Researchers will compare the effect of the Modified Sleeper-Stretch in the elasticity of the posterior and posteroinferior glenohumeral capsule in individuals with history of shoulder pain applying the technique on the affected shoulder and comparing with the healthy shoulder. In healthy individuals the intervention will be made on a randomly assigned shoulder and the effect will be compared to the non-interventional shoulder. Finally, a comparison between groups will be made considering only the intervention shoulder to see if there are differences in the effect amongst healthy and affected individuals.

Participants will be asked to follow a self-administered Modified Sleeper-Stretch program consisting of the execution of the stretch three times, for thirty seconds each time, with thirty seconds between stretches, daily, for twenty-eight days.

DETAILED DESCRIPTION:
Non-specific shoulder pain is the third most frequent among musculoskeletal pains. It causes functional limitation that can lead to capsular stiffness and restriction of movement. Interventions aimed at reducing posterior capsule stiffness may improve the symptoms of painful shoulder. Modified Sleeper-Stretch is credited with the ability to decrease posterior shoulder stiffness. Shear-wave elastography is an imaging technique capable of quantifying the stiffness of the posterior capsule of the shoulder.

The objective of this study is to determine the effect of a stretching program using Modified Sleeper-Stretch on the elasticity of the posterior and posteroinferior capsule of the glenohumeral joint in adult population with and without a history of non-specific shoulder pain, using shear-wave elastography.

A quasi-experimental pre-post study will be conducted over two experimental groups of 32 subjects each. The intervention will involve following a self-stretching program of the posterior region of the shoulder using modified sleeper-stretch for 28 days. The study subjects will be adult individuals with a history of non-specific shoulder pain in the first group and no history of shoulder pain in the second. The first group will follow the program on the affected shoulder, the second on a randomly assigned shoulder. The elasticity of the posterior and posteroinferior glenohumeral capsule will be measured by shear-wave elastography in both shoulders at the beginning of the intervention, at its completion and four weeks after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with clinical history of nonspecific shoulder pain on a single shoulder, who had GIRD of 15º or more, asymptomatic for more than one month and less than one year.
* Male or female with no history of shoulder pain.
* Age between 18 and 59 years.

Exclusion Criteria:

* Glenohumeral osteoarthritis.
* Labrum lesion, Bankart or Hill-Sachs lesion.
* Posterior instability of any of the shoulders.
* Evidence of joint hypermobility as defined by a Beighton Scale score greater or equal to 6.
* Rotator cuff tear.
* Fracture or surgery in the cervical region or in any of the upper limbs, except shoulders, if less than a year has passed since the episode.
* History of surgical intervention in any of the shoulders.
* Tumor growth in the shoulder region.
* Neuromuscular injuries with shoulder muscles motor involvement (myasthenia, spinal cord injury, spastic contracture, paresis).
* Inflammatory diseases (rheumatoid arthritis, psoriatic arthritis) affecting the shoulder region in state of outbreak.
* Metabolic or systemic diseases with potential to modify tissue elastic capacity.
* Diseases or injuries with contraindication to mobilization or physical exercise of the shoulder region.
* Inability to perform the stretch due to pain.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Posterior glenohumeral capsule elasticity | Day 1 (twice), day 28 (twice), day 56 (once)
  Elasticity of posterior glenohumeral capsule as determined by quantitative shear-wave elastography
Posteroinferior glenohumeral capsule elasticity | Day 1 (twice), day 28 (twice), day 56 (once)
  Elasticity of posteroinferior glenohumeral capsule as determined by quantitative shear-wave elastography

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Ramirez-Llano, PT, Principal Investigator — Member of the department
Locations (1):
- Departamento de Enfermería y Fisioterapia, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
All the information obtained in the study will be only published on a statistical basis. Only the principial investigator of the study will be able to associate information of the study with any individual participant.

REFERENCES:
- [Background] Jacome-Lopez R, Tejada-Gallego J, Silberberg JM, Garcia-Sanz F, Garcia-Muro-San Jose F. Glenohumeral internal rotation deficit in general population with shoulder pain: A descriptive observational study. Medicine (Baltimore). 2023 Dec 15;102(50):e36551. doi: 10.1097/MD.0000000000036551. PMID 38115341
- [Background] Rosa DP, Borstad JD, Ferreira JK, Gava V, Santos RV, Camargo PR. Comparison of specific and non-specific treatment approaches for individuals with posterior capsule tightness and shoulder impingement symptoms: A randomized controlled trial. Braz J Phys Ther. 2021 Sep-Oct;25(5):648-658. doi: 10.1016/j.bjpt.2021.04.003. Epub 2021 May 4. PMID 34001426
- [Background] Borstad JD, Dashottar A. Quantifying strain on posterior shoulder tissues during 5 simulated clinical tests: a cadaver study. J Orthop Sports Phys Ther. 2011 Feb;41(2):90-9. doi: 10.2519/jospt.2011.3357. Epub 2010 Nov 10. PMID 21169717
- [Background] Laudner KG, Sipes RC, Wilson JT. The acute effects of sleeper stretches on shoulder range of motion. J Athl Train. 2008 Jul-Aug;43(4):359-63. doi: 10.4085/1062-6050-43.4.359. PMID 18668168
- [Background] Wilk KE, Hooks TR, Macrina LC. The modified sleeper stretch and modified cross-body stretch to increase shoulder internal rotation range of motion in the overhead throwing athlete. J Orthop Sports Phys Ther. 2013 Dec;43(12):891-4. doi: 10.2519/jospt.2013.4990. Epub 2013 Oct 30. PMID 24175603
- [Background] Mine K, Nakayama T, Milanese S, Grimmer K. Effectiveness of Stretching on Posterior Shoulder Tightness and Glenohumeral Internal-Rotation Deficit: A Systematic Review of Randomized Controlled Trials. J Sport Rehabil. 2017 Jul;26(4):294-305. doi: 10.1123/jsr.2015-0172. Epub 2016 Aug 24. PMID 27632891
- [Background] Izumi T, Aoki M, Muraki T, Hidaka E, Miyamoto S. Stretching positions for the posterior capsule of the glenohumeral joint: strain measurement using cadaver specimens. Am J Sports Med. 2008 Oct;36(10):2014-22. doi: 10.1177/0363546508318196. Epub 2008 Jun 20. PMID 18567716
- [Background] McClure P, Balaicuis J, Heiland D, Broersma ME, Thorndike CK, Wood A. A randomized controlled comparison of stretching procedures for posterior shoulder tightness. J Orthop Sports Phys Ther. 2007 Mar;37(3):108-14. doi: 10.2519/jospt.2007.2337. PMID 17416125
- [Background] Yamauchi T, Hasegawa S, Nakamura M, Nishishita S, Yanase K, Fujita K, Umehara J, Ji X, Ibuki S, Ichihashi N. Effects of two stretching methods on shoulder range of motion and muscle stiffness in baseball players with posterior shoulder tightness: a randomized controlled trial. J Shoulder Elbow Surg. 2016 Sep;25(9):1395-403. doi: 10.1016/j.jse.2016.04.025. Epub 2016 Jul 27. PMID 27475455
- [Background] Tawfik A, Toci GR, Sirch F, Gibbs B, Conte E, Fletcher D, Hornstein J, Aland C. The Effects of Sleeper and Superman Stretches on Time-Zero Shoulder Range of Motion in Collegiate Athletes. Cureus. 2022 Feb 25;14(2):e22600. doi: 10.7759/cureus.22600. eCollection 2022 Feb. PMID 35371739
- [Background] Chepeha JC, Magee DJ, Bouliane M, Sheps D, Beaupre L. Effectiveness of a Posterior Shoulder Stretching Program on University-Level Overhead Athletes: Randomized Controlled Trial. Clin J Sport Med. 2018 Mar;28(2):146-152. doi: 10.1097/JSM.0000000000000434. PMID 28731885
- [Background] Takenaga T, Sugimoto K, Goto H, Nozaki M, Fukuyoshi M, Tsuchiya A, Murase A, Ono T, Otsuka T. Posterior Shoulder Capsules Are Thicker and Stiffer in the Throwing Shoulders of Healthy College Baseball Players: A Quantitative Assessment Using Shear-Wave Ultrasound Elastography. Am J Sports Med. 2015 Dec;43(12):2935-42. doi: 10.1177/0363546515608476. Epub 2015 Oct 15. PMID 26473012
- [Background] Iida N, Taniguchi K, Watanabe K, Miyamoto H, Taniguchi T, Fujimiya M, Katayose M. Relationship between shear modulus and passive tension of the posterior shoulder capsule using ultrasound shear wave elastography: A cadaveric study. J Biomech. 2020 Jan 23;99:109498. doi: 10.1016/j.jbiomech.2019.109498. Epub 2019 Nov 9. PMID 31735360
- [Background] Iida N, Taniguchi K, Watanabe K, Miyamoto H, Taniguchi T, Teramoto A, Katayose M. Effective stretching positions for the posterior shoulder capsule as determined by shear wave elastography. J Shoulder Elbow Surg. 2021 May;30(5):1186-1195. doi: 10.1016/j.jse.2020.08.021. Epub 2020 Sep 9. PMID 32919046